CLINICAL TRIAL: NCT04823741
Title: Molecular, Pathologic Intra Tumoral Heterogeneity in Malignant Pleural Mesothelioma
Acronym: SCITH-MESO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0997; 2021-A00748-33 (Other: ID-RCB)
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Mesothelioma, Malignant; Gene Abnormality; Pleural Mesothelioma
Keywords: malignant pleural mesothelioma; intra tumoral heterogeneity; genetic abnormalities
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — pleural samples of malignant pleural mesothelioma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PLEURAL BIOCOLLECTION OF MALIGNANT PLEURAL MESOTHELIOMA: All patient with suspected malignant pleural mesothelioma requiring surgical biopsy after validation in oncologic multidisciplinary board will be included. During a standardized routine procedure of pleural biopsy by mean of general anesthesia and video thoracoscopic approach, 3 - 5 biopsies are realized. During this procedure, blood samples are collected and a piece of biopsy will be used for the constitution of a specific bio collection in the CRB (centre de ressources biologiques).
  Interventions: Genetic: PLEURAL BIOCOLLECTION OF MALIGNANT PLEURAL MESOTHELIOMA

INTERVENTIONS:
Genetic: PLEURAL BIOCOLLECTION OF MALIGNANT PLEURAL MESOTHELIOMA — All patient with suspected malignant pleural mesothelioma requiring surgical biopsy after validation in oncologic multidisciplinary board will be included. During a standardized routine procedure of pleural biopsy by mean of general anesthesia and video thoracoscopic approach, 3 - 5 biopsies are realized. During this procedure, blood samples are collected and a piece of biopsy will be used for the constitution of a specific bio collection in the CRB (centre de ressources biologiques).

SUMMARY:
Malignant pleural mesothelioma (MPM) is a rare pleural cancer, which could be primary or secondary to an asbestos exposure. To enhance our knowledge of this rare disease, an exploration of genetic and tumor mechanism is mandatory. One of the principal difficulty is to harvest sufficient tumour pieces to perform multi-omics analysis. The goal of the SCITH-MESO study is to harvest larges pieces of tumour during a routine surgical procedure of MPM diagnosis by mean of pleural biopsies during VATS surgery. Operating samples will increase a tissue bank collection (CRB).

ELIGIBILITY:
Inclusion Criteria:

* age >18
* suspected MPM requiring VATS biopsy after multidisciplinary oncologic board validation
* patient able to understand study objectives and able to give an informed consent
* patient affiliated to an healthcare society.

Exclusion Criteria:

* pregnancy
* mental disease, psychiatric disorder
* patient under protection regimen

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patient with suspected malignant pleural mesothelioma requiring surgical biopsy for diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2026-02-11 (Estimated); Study Completion 2026-02-11 (Estimated)

PRIMARY OUTCOMES:
For patients with MPM, blood samples are collected and a piece of biopsy will be used for the constitution of a specific bio collection in the CRB (centre de ressources biologiques). | day 1 (day of chirurgie)
  For patients with MPM, blood samples are collected and a piece of biopsy will be used for the constitution of a specific bio collection in the CRB (centre de ressources biologiques).

CONTACTS AND LOCATIONS:
Locations (1):
- Département de chirurgie thoracique, Bron, France